CLINICAL TRIAL: NCT03058601
Title: Health Outcomes of Patients With Acute Coronary Syndromes Prescribed Ticagrelor in UK Primary Care: a Retrospective Cohort Study
Brief Title: Outcomes in UK ACS Patients Prescribed Ticagrelor
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5130R00027; EUPAS17107 (Registry Identifier: ENCePP)
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Cohort study using data from Clinical Practice Research Datalink (CPRD). The study cohort includes all patients who received at least one prescription for ticagrelor for the first time between December 2010 and March 2015, following ACS. Patient baseline characteristics will be described: (Age, Gender, Body Mass Index, Smoking status, Sociodemographic status), type of ACS and interventions, CV history and comorbidities, bleeding and respiratory history.

The following outcomes will be examined: Incidence of vascular events (composite MI, Stroke, vascular death, specific vascular event and all cause death), incidence of bleeding and incidence of dysponea. Time to event for vascular events, bleeding and dyspnoea.

ELIGIBILITY:
Inclusion Criteria:

* First prescription (index date) for ticagrelor between Dec 2010 and Mar 2015
* At least 12 months history in database prior to first ticagrelor prescription
* Linkage to Hospital Episode Statistics (HES)
* Acute Coronary Syndrome (ACS) event in the three months prior to and including the index date

Exclusion Criteria:

Primary care prescription for clopidogrel or prasugrel between the ACS date and the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients prescribed ticagrelor in primary care, following Acute Cornoary Syndrome (ACS), for the first time (Dec 2010 - Mar 2015) in Cliniical Practice Research Datalink primary care data and followed for up to 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of composite outcome of myocardial infarction (MI), Stroke or death from vascular causes in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months
Incidence of myocardial infarction (MI) in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months
Incidence of all cause death in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months
Incidence of stroke in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months
Incidence of vascular death in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months
Time to event for composite outcome of myocardial infarction (MI), Stroke or death from vascular causes in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months
Time to event for myocardial infarction (MI) in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months
Time to event for all cause death in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months
Time to event for stroke in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months
Time to event for vascular death in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months

SECONDARY OUTCOMES:
Incidence of bleeding in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months
Incidence of dyspnoea in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months
Time to event for bleeding in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months
Time to event for dyspnoea in patients treated with ticagrelor in primary care following Acute Coronary Syndrome (ACS) | From index date up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Luton, United Kingdom

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14606&filename=Synopsis_of_Study%20Report_D5130R00027_Redacted.pdf